CLINICAL TRIAL: NCT01157117
Title: Oral Immunotherapy Combined With Humanized Monoclonal Anti-IgE Antibody Xolair® (Omalizumab)in the Treatment of Cow's Milk Allergy
Brief Title: OIT and Xolair® (Omalizumab) in Cow's Milk Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hugh A Sampson, MD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Hugh A Sampson, MD, Dean for Translational Biomedical Sciences, Director, Jaffe Food Allergy Institute, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT AADCRC-MSSM-01; U19AI044236 (NIH)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Milk Allergy
Keywords: food allergy
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity | interventions — Omalizumab; Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Omalizumab/milk OIT (Experimental): Participants receive blinded omalizumab injections every 2 to 4 weeks through Month 16 and unblinded omalizumab injections thereafter until the Month 28 desensitization oral food challenge (OFC). Participants ingest milk powder daily starting at Month 4 with a dose of 0.07 mg milk protein and escalate for 22 to 40 weeks until reaching the maintenance dose of 3.84 g milk protein (minimum required maintenance dose is 520 mg milk protein). At Month 28, participants complete a 10g milk OFC and discontinue omalizumab injections. If they fail the OFC they permanently discontinue ingestion of the milk powder; if they pass the OFC they continue ingestion of the maintenance dose of milk powder through Month 30 and then discontinue it.
  Interventions: Biological: Omalizumab; Drug: Milk powder
- Placebo for omalizumab/milk OIT (Placebo Comparator): Participants receive blinded placebo for omalizumab injections every 2 to 4 weeks through Month 16; after unblinding the injections are discontinued. Participants ingest milk powder daily starting at Month 4 with a dose of 0.07 mg milk protein and escalate for 22 to 40 weeks until reaching the maintenance dose of 3.84 g milk protein (minimum required maintenance dose is 520 mg milk protein). At Month 28, participants complete a 10g milk oral food challenge (OFC); if they fail the OFC they permanently discontinue ingestion of the milk powder; if they pass the OFC they continue ingestion of the maintenance dose of milk powder through Month 30 and then discontinue it.
  Interventions: Biological: Placebo for omalizumab; Drug: Milk powder
- Untreated control (No Intervention): Participants did not receive any study intervention but provided regular blood draws at specific study time points to allow mechanistic comparisons with the participants in the other two groups who did receive study intervention.

INTERVENTIONS:
Biological: Placebo for omalizumab — Placebo for omalizumab is injected subcutaneously every 2-4 weeks for 16 months at a volume designed to match that of the verum treatment group (determined by the participant's IgE level and weight).
  Other Names: Placebo for Xolair
  Arms: Placebo for omalizumab/milk OIT
Biological: Omalizumab — Omalizumab is injected subcutaneously every 2-4 weeks for 28 months at a dose determined by the participants IgE level and weight.
  Other Names: Xolair
  Arms: Omalizumab/milk OIT
Drug: Milk powder — Milk powder is ingested orally at a dosage of up to 3.84 grams of of milk protein daily from Month 4 through Month 28 if the Month 28 10 g milk OFC is failed, and through Month 30 if the Month 28 10 g milk OFC is passed.
  Arms: Omalizumab/milk OIT; Placebo for omalizumab/milk OIT

SUMMARY:
Food allergy affects up to 4% of the U.S. population and is most common in young children. Milk allergy is the most common cause of food allergy in infants and young children, and usually develops in the first year of life. There is no treatment for food allergy and the current standard of care for milk-allergic individuals is the avoidance of milk-containing products. Research is underway to identify potential therapeutic strategies to reduce or eliminate the adverse effects experienced by milk-allergic individuals when they consume milk-containing products.

Several studies have suggested that milk-allergic children who receive milk protein oral immunotherapy (OIT) may become desensitized to milk, resulting in short term protection against accidental ingestion of milk products. However, these children did not develop "tolerance," which is long term protection even after milk immunotherapy is stopped. A potential strategy to induce tolerance to milk uses milk in combination with Xolair® (omalizumab). Xolair consists of anti-IgE molecules that attach to IgE, the major antibody involved in allergic reactions. The goal of this clinical trial is to see whether Xolair® in combination with milk protein OIT is safer and more effective than OIT alone in inducing tolerance to milk and milk products. Participants will be administered a double blind, placebo controlled milk challenge at various time points in the study. If desensitization is achieved participants will be tested for tolerance at a certain time point after stopping treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or parent/ legal guardian must be able to understand and provide written informed consent
* Written or verbal assent from all study subjects less than 18 years (per site Institutional Review Board (IRB) regulations)
* 7 to 35 years of age; any gender; any racial and ethnic origin
* No known contraindications to therapy using oral immunotherapy with milk protein or Xolair® (omalizumab)
* All female subjects of childbearing potential must have a negative pregnancy test upon study entry
* All treated females of childbearing potential must agree to use FDA approved methods of birth control for the duration of the study

Active Treatment Subjects:

* Cow's milk allergy confirmed by a positive double-blind placebo controlled milk challenge (DBPCMC) to a dose of less than 2 g of milk protein within the past 6 months
* A skin prick test positive to milk (diameter of wheal >= 3.0 mm) OR detectable serum milk specific Immunoglobulin E (IgE) level within the previous 12 months (UniCAP > = 0.35 kUA/L (allergen-equivalent kilounits per liter))

Control Subjects:

• A skin prick test positive to milk (diameter of wheal >= 10.0 mm) OR detectable serum milk specific IgE level within the previous 12 months (UniCAP >= 15 kUA/L)

Exclusion Criteria:

* A history of life-threatening anaphylaxis to milk (involving hypotension or requiring mechanical ventilation)
* Known allergy to any components of the placebo for Xolair®
* Chronic disease other than asthma, atopic dermatitis, or allergic rhinitis requiring therapy (e.g., heart disease, diabetes)
* Use of β-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB), or calcium channel blockers
* Severe asthma
* Mild or moderate asthma with any of the following criteria met:

  * Forced expiratory volume in the first second (FEV1) < 80% with or without controller medications
  * Inhaled corticosteroids (ICS) dosing of >500 mcg daily fluticasone (or equivalent inhaled corticosteroids based on NHLBI dosing chart)
  * history of daily oral steroid dosing for >1 month during the past year
  * burst oral steroid course in the past 6 months
  * more than one burst oral steroid course in the past year
  * more than one hospitalization in the past year for asthma, or
  * more than one ER visit in the past 6 months for asthma
* Baseline spirometry (or peak flow rate (PFR) if unable to perform spirometry) result of FEV1<80%
* Pregnancy or lactation. All females of child-bearing age will undergo pregnancy testing. All treated females will confirm compliance to appropriate birth control measures throughout the course of the study;
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Subject is on a buildup phase of standard subcutaneous immunotherapy for inhalant allergens (may be enrolled on maintenance dose);
* Use of Xolair® (omalizumab) or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual immunotherapy) or immunomodulator therapy (not including corticosteroids) or biologic therapy within the past year
* Inability to discontinue antihistamines for 5 half-lives prior to routine study tests (DBPCMC or endpoint titration tests)
* Known sensitivity to Xolair® (omalizumab) or to the class of study drugs
* Baseline serum total IgE over 1,300 IU/mL or body weight more than 150 kg, or subjects with weight-IgE combination that yields a dose requirement greater than 750 mg (due to limitations of Xolair® (omalizumab) dosing)
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements
* Inability or unwillingness of a subject to give written informed consent or comply with study protocol
* Use of investigational drugs within 90 days of participation
* Other contraindications to milk oral immunotherapy or Xolair® (omalizumab)
* Recipient of any licensed or investigational live attenuated vaccine(s) within 2 months of enrollment
* Families who do not speak English
* Systemic steroids oral, intramuscular (IM), or IV for indications other than asthma for greater than 3 weeks in the past 6 months

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2010-08; Primary Completion 2015-01 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A. Sampson, M.D., Study Chair — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Result] Wood RA, Kim JS, Lindblad R, Nadeau K, Henning AK, Dawson P, Plaut M, Sampson HA. A randomized, double-blind, placebo-controlled study of omalizumab combined with oral immunotherapy for the treatment of cow's milk allergy. J Allergy Clin Immunol. 2016 Apr;137(4):1103-1110.e11. doi: 10.1016/j.jaci.2015.10.005. Epub 2015 Nov 12. PMID 26581915
- [Derived] Noone S, Ross J, Sampson HA, Wang J. Epinephrine use in positive oral food challenges performed as a screening test for food allergy therapy trials. J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):424-8. doi: 10.1016/j.jaip.2014.10.008. Epub 2015 Jan 13. PMID 25609353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at three university-based medical centers in the United States (Mount Sinai, Johns Hopkins University, Stanford University) beginning in October 2010. Accrual of randomized participants was completed in April 2012 and of untreated controls was completed in August 2012.
Groups:
- Omalizumab/Milk OIT: Participants receive blinded omalizumab injections every 2 to 4 weeks through Month 16 and unblinded omalizumab injections thereafter until the Month 28 desensitization OFC. Participants ingest milk powder daily starting at Month 4 with a dose of 0.07 mg milk protein and escalate for 22 to 40 weeks until reaching the maintenance dose of 3.84 g milk protein (minimum required maintenance dose is 520 mg milk protein). At Month 28 participants complete a 10g milk OFC and discontinue omalizumab injections. If they fail the OFC they permanently discontinue ingestion of the milk powder; if they pass the OFC they continue ingestion of the maintenance dose of milk powder through Month 30 and then discontinue it.
- Placebo for Omalizumab/Milk OIT: Participants receive blinded placebo for omalizumab injections every 2 to 4 weeks through Month 16; after unblinding the injections are discontinued. Participants ingest milk powder daily starting at Month 4 with a dose of 0.07 mg milk protein and escalate for 22 to 40 weeks until reaching the maintenance dose of 3.84 g milk protein (minimum required maintenance dose is 520 mg milk protein). At Month 28 participants complete a 10g milk OFC; if they fail the OFC they permanently discontinue ingestion of the milk powder; if they pass the OFC they continue ingestion of the maintenance dose of milk powder through Month 30 and then discontinue it.
Period: Overall Study
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Started | 28 | 29 | 20
Began Omalizumab or Placebo Dosing | 27 | 28 | 0
Began Milk OIT Dosing at Month 4 | 27 | 28 | 0
Reached Milk OIT Maintenance Dosing | 26 | 26 | 0
Unblinded at Month 16 | 26 | 26 | 0
Completed Month 28 Desensitization OFC | 26 | 24 | 0
Discontinued Milk OIT at Month 30 | 24 | 20 | 0
Completed Month 32 Tolerance OFC | 24 | 20 | 0
Completed Final Month 38 Study Visit | 19 | 18 | 3
Completed | 19 (Completed final study visit at Month 38, 6 months after final Month 32 OFC.) | 18 (Completed final study visit at Month 38, 6 months after final Month 32 OFC.) | 5 (Completed final study visit at Month 38, 6 months after final Month 32 OFC.)
Not Completed | 9 | 11 | 15
Not completed — Dosing Symptoms | 0 | 4 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Unknown (Pending Final Form Submission) | 4 | 5 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control | Total
Number analyzed (Participants) | 28 | 29 | 20 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 27 | 20 | 73
  Between 18 and 65 years | 2 | 2 | 0 | 4
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 5 | 22
  Male | 20 | 20 | 15 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino origin | 0 | 2 | 0 | 2
  Non-Hispanic or non-Latino origin | 28 | 27 | 20 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4 | 3 | 2 | 9
  Black/African American | 1 | 0 | 0 | 1
  White | 23 | 26 | 18 | 67
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 20 | 77
Age [Mean (Standard Deviation); unit: years] | 12.6 (4.1) | 11.5 (5.6) | 11.3 (2.9) | 11.8 (4.5)
Atopic Dermatitis Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Atopic Dermatitis Total Score is scored on a 10 point scale of 0 to 9 where a higher score indicates increasing severity of atopic dermatitis. This score is a combination of three scores that range from 0 to 3 in the following areas: body surface area score, disease course, and disease intensity. Note: These data were only available for 12 of the 20 Untreated Control participants.
  Scores on a scale | 0.3 (0.9) | 0.5 (1.5) | 1.0 (2.3) | 0.5 (1.5)
Total IgE [Mean (Standard Deviation); unit: kU/L] — Total amount of serum immunoglobulin E (IgE).
  kU/L | 683.1 (658.9) | 686.6 (565.7) | 878.8 (824.3) | 735.2 (670.3)
Milk IgE [Mean (Standard Deviation); unit: kUA/L] — Amount of serum milk-specific immunoglobulin E (IgE). Individuals with a milk IgE of <0.35 kUA/L (allergen-equivalent kilounits per liter) are considered not to be sensitized to milk.
  kUA/L | 52.2 (47.4) | 57.9 (55.5) | 72.4 (63.9) | 59.6 (54.9)
Milk Skin Prick Test Score [Mean (Standard Deviation); unit: mm] — This score is calculated by subtracting the size of the saline wheal (in mm) from the size of the milk wheal (in mm) observed for a skin prick test. Individuals with a milk skin prick test score of < 3 mm are considered to have a negative result.
  mm | 8.9 (3.3) | 9.0 (3.2) | NA (NA) — Data were not collected for this group. | 8.9 (3.2)
Age at Initial Milk Allergic Reaction [Mean (Standard Deviation); unit: years] — Age in years at the participant's first milk allergic reaction. Note: These data were only available for 14 of the 28 Omalizumab/Milk OIT participants, 19 of the 29 Placebo for Omalizumab/Milk OIT participants, and 14 of the 20 Untreated Control participants.
  years | 0.9 (1.8) | 0.5 (0.5) | 0.9 (0.8) | 0.7 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in the Xolair® (Omalizumab) Group vs. Placebo Group Developing Clinical Tolerance to Milk
Description: Tolerance Assessment: Participants who successfully consumed without dose-limiting symptoms 10,000 mg of milk protein during a double-blind placebo-controlled oral food challenge were then given an open feeding of milk and those who successfully consumed the open feeding were counted as successes.
Time Frame: Month 32 which is 8 weeks following the discontinuation of milk OIT for both groups and 4 months after discontinuation of omalizumab for the omalizumab group
Population: The intention to treat (ITT) population was used which included all subjects randomized to double-blind treatment.
Measure: Number; unit: Percent of participants
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 28 | 29
Percent of participants | 46.4 | 34.5
Statistical Analysis 1: Comparison: Omalizumab/Milk OIT vs Placebo for Omalizumab/Milk OIT; Number of participants who successfully consumed 10,000 mg of milk protein followed by an open feeding of milk was compared using Fisher's Exact test with the null hypothesis that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.42, Fisher Exact — No adjustments were made to the p-value; The a priori threshold for statistical significance is 0.05; Risk Difference (RD) = 12.0, 95% CI 2-sided [-13.4 to 37.3]

2. Secondary Outcome: Incidence of Dosing Reactions to Milk OIT During the Escalation Phase
Description: Any reaction to daily milk OIT dosing recorded by the participant during the Escalation Phase.
Time Frame: Baseline to completion of Escalation Phase at 22 to 40 weeks
Population: Participants who received any milk OIT dosing during the Escalation Phase.
Measure: Number; unit: percentage of participants
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 27 | 28
percentage of participants | 81.5 | 96.4

3. Secondary Outcome: Incidence of Dosing Reactions to Milk OIT During the Maintenance Phase
Description: Any reaction to daily milk OIT dosing recorded by the participant during the Maintenance Phase.
Time Frame: After completion of Escalation Phase at 22 to 40 weeks, the Maintenance Phase lasted up to Month 30
Population: Participants who received milk OIT dosing during the Maintenance Phase.
Measure: Number; unit: percentage of participants
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 26 | 26
percentage of participants | 46.2 | 96.2

4. Secondary Outcome: Incidence of Severe Hypersensitivity Reactions to Milk OIT
Description: Participants who had a change in mental status or hypotension as a milk OIT dosing symptom were counted as having a severe hypersensitivity reaction.
Time Frame: Through completion of milk OIT dosing (at Month 28 if failed desensitization OFC, at Month 30 if passed desensitization OFC)
Population: Participants who received milk OIT dosing.
Measure: Number; unit: percentage of participants
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 27 | 28
percentage of participants | 0 | 0

5. Secondary Outcome: Maximum Tolerated Dose of Milk Oral Immunotherapy (OIT)
Description: Maximum tolerated dose of milk OIT is the highest dose of milk powder the participant was able to consume for at least 14 consecutive days.
Time Frame: Baseline to completion of Escalation Phase at 22 to 40 weeks
Population: Participants who received any milk OIT dosing
Measure: Mean (Standard Deviation); unit: mg milk powder
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 27 | 28
mg milk powder | 9941.7 (2692.9) | 9174.0 (3344.6)

6. Secondary Outcome: Percentage of Participants in the Xolair® (Omalizumab) Group vs. Placebo Group Developing Desensitization to Milk
Description: Desensitization Assessment: Participants who successfully consumed without dose-limiting symptoms 10,000 mg of milk protein during a double-blind placebo-controlled oral food challenge were counted as successes.
Time Frame: Month 28
Population: Participants who received any study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 27 | 28
percentage of participants | 88.9 | 71.4

7. Secondary Outcome: Time to Maximum Tolerated Dose
Description: Time to reach the maximum tolerated dose (MTD) of milk oral immunotherapy (OIT); MTD is the highest dose of milk powder the participant was able to consume for at least 14 consecutive days.
Time Frame: Baseline to completion of Escalation Phase at 22 to 40 weeks
Population: Time to maximum tolerated dose could not be calculated because the maximum dose for the protocol was changed part way through the study after some subjects had already reached the maximum dose.
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline to Month 32 in Area Under the Curve for Milk Endpoint Titration Prick Skin Test
Description: A milk endpoint titration is a prick skin test using 5 serial 10-fold dilutions of milk which include 1:20 wt/vol, 1:200 wt/vol, 1:2,000 wt/vol, 1:20,000 wt/vol and 1:200,000 wt/vol. The score for each of these dilutions is calculated by subtracting the diameter of the saline control wheal from the diameter of the milk wheal (in millimeters). The area under the curve is calculated by adding together the scores from all 5 milk dilutions creating a composite score.
Time Frame: Month 32
Population: All randomized participants who had not withdrawn from the study and came to the clinic for their Month 32 visit were assessed.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT
Number analyzed (Participants) | 25 | 22
units on a scale | -12.5 [-32.0 to 3.0] | -15.3 [-45.0 to -1.5]

9. Secondary Outcome: Change From Baseline to Month 32 in Antigen-specific Immunoglobulin E (IgE)
Description: The level of milk IgE in plasma as well as the IgE levels of 2 milk proteins, casein and beta-lactoglobulin, were measured. The value for each participant was subtracted from the value for that participant at baseline. Month 32 was the last visit on treatment.
Time Frame: Month 32
Population: All randomized participants and untreated controls who had not withdrawn from the study, came to the clinic for their Month 32 visit, and for whom valid results were reported.
Measure: Median (Full Range); unit: kUA/L
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 25 | 22 | 6
kUA/L
  Change in Milk IgE | -9.8 [-134.2 to 50.5] | -16.9 [-121.7 to 200.0] | 0.8 [-78.4 to 103.4]
  Change in Casein IgE | -6.2 [-194.1 to 596.0] | -27.7 [-170.6 to 69.0] | 3.5 [-76.1 to 177.2]
  Change in Beta-lactoglobulin IgE | -1.7 [-72.5 to 59.1] | -2.9 [-129.5 to 41.6] | 7.2 [-33.7 to 41.7]

10. Secondary Outcome: Change From Baseline to Month 32 in Antigen-specific Immunoglobulin G4 (IgG4)
Description: Casein and beta-lactoglobulin milk proteins IgG4 levels were measured in plasma. The value for each participant was subtracted from the value for that participant at baseline. Month 32 was the last visit on treatment.
Time Frame: Month 32
Population: as for outcome 9
Measure: Median (Full Range); unit: mgA/L
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 25 | 22 | 6
mgA/L
  Change in Casein IgG4 | 17.3 [0.2 to 57.2] | 13.5 [-0.2 to 47.4] | 0.1 [-0.3 to 60.4]
  Change in Beta-lactoglobulin IgG4 | 24.9 [-0.1 to 58.7] | 20.8 [-0.1 to 62.3] | -0.02 [-1.3 to 52.5]

11. Secondary Outcome: Change From Baseline to Month 38 in Antigen-specific Immunoglobulin E (IgE)
Description: The level of milk IgE in plasma as well as the IgE levels of 2 milk proteins, casein and beta-lactoglobulin, were measured. The value for each participant was subtracted from the value for that participant at baseline. Month 38 was 6 months after treatment ended at Month 32.
Time Frame: Month 38
Population: All randomized participants and untreated controls who had not withdrawn from the study, came to the clinic for their Month 38 visit, and for whom valid results were reported.
Measure: Median (Full Range); unit: kUA/L
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 18 | 18 | 5
kUA/L
  Change in Milk IgE | -25.1 [-135.6 to 37.0] | -15.8 [-147.5 to 18.1] | -1.0 [-8.3 to 95.4]
  Change in Casein IgE | -14.9 [-194.8 to 58.0] | -34.8 [-189.5 to 7.4] | 1.6 [-0.6 to 71.2]
  Change in Beta-lactoglobulin IgE | -2.7 [-73.8 to 68.1] | -2.6 [-139.2 to 91.1] | 1.9 [-13.1 to 28.0]

12. Secondary Outcome: Change From Baseline to Month 38 in Antigen-specific Immunoglobulin G4 (IgG4)
Description: Casein and beta-lactoglobulin milk proteins IgG4 levels were measured in plasma. The value for each participant was subtracted from the value for that participant at baseline. Month 38 was 6 months after treatment ended at Month 32.
Time Frame: Month 38
Population: as for outcome 11
Measure: Median (Full Range); unit: mgA/L
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 18 | 18 | 5
mgA/L
  Change in Casein IgG4 | 44.9 [0.6 to 100.3] | 21.0 [-1.5 to 56.5] | 0.4 [-0.6 to 16.6]
  Change in Beta-lactoglobulin IgG4 | 23.8 [0.1 to 121.5] | 25.6 [-2.6 to 125.0] | -0.02 [-0.7 to 0.3]

13. Secondary Outcome: Change in Percent of Cells Positive for Cluster of Differentiation 63 (CD63) at Month 32 in Basophils Stimulated by Milk
Description: Basophil cells isolated from blood using flow cytometry were stimulated with 5 different levels of milk and the percent of basophil cells that were CD63 positive was measured. The value for each participant obtained at Month 32 was subtracted from the value for that participant at baseline. The 5 different levels of milk stimulant were: 10 µg/mL, 1 µg/mL , 0.1 µg/mL , 0.01 µg/mL , and 0.001 µg/mL. Month 32 was the last visit on treatment.
Time Frame: Month 32
Population: as for outcome 9
Measure: Median (Full Range); unit: percentage of CD63+ basophils
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 21 | 19 | 5
percentage of CD63+ basophils
  Change in %CD63+ for 10 µg/mL stimulant | 11.1 [-19.8 to 81.2] | 8.7 [-61.4 to 76.0] | 13.0 [10.3 to 25.5]
  Change in %CD63+ for 1 µg/mL stimulant | 7.5 [-37.3 to 74.2] | 0.6 [-56.6 to 85.2] | 6.9 [-2.6 to 40.9]
  Change in %CD63+ for 0.1 µg/mL stimulant | -11.8 [-57.3 to 34.2] | -5.5 [-53.2 to 79.1] | 15.9 [-7.3 to 45.9]
  Change in %CD63+ for 0.01 µg/mL stimulant | -6.5 [-47.5 to 23.2] | -3.8 [-59.2 to 87.6] | 26.2 [-4.7 to 35.5]
  Change in %CD63+ for 0.001 µg/mL stimulant | -1.3 [-41.5 to 19.1] | -1.2 [-44.0 to 85.5] | 1.9 [-1.7 to 7.5]

14. Secondary Outcome: Change in Percent of Cells Positive for Cluster of Differentiation 63 (CD63) at Month 38 in Basophils Stimulated by Milk
Description: Basophil cells isolated from blood using flow cytometry were stimulated with 5 different levels of milk and the percent of basophil cells that were CD63 positive was measured. The value for each participant obtained at Month 38 was subtracted from the value for that participant at baseline. The 5 different levels of milk stimulant were: 10 µg/mL, 1 µg/mL , 0.1 µg/mL , 0.01 µg/mL , and 0.001 µg/mL. Month 38 was 6 months after treatment ended at Month 32.
Time Frame: Month 38
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of CD63+ basophils
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Number analyzed (Participants) | 19 | 18 | 5
percentage of CD63+ basophils
  Change in %CD63+ for 10 µg/mL stimulant | -9.2 [-59.3 to 56.6] | -11.7 [-72.9 to 46.1] | 26.7 [14.0 to 53.0]
  Change in %CD63+ for 1 µg/mL stimulant | -8.2 [-53.1 to 17.2] | -9.5 [-57.5 to 57.7] | 29.5 [-0.2 to 37.8]
  Change in %CD63+ for 0.1 µg/mL stimulant | -18.6 [-59.4 to 1.8] | -21.6 [-63.0 to 0.0] | 28.6 [17.2 to 42.2]
  Change in %CD63+ for 0.01 µg/mL stimulant | -10.2 [-61.9 to 0.5] | -7.8 [-64.5 to 8.5] | 8.4 [-10.1 to 36.2]
  Change in %CD63+ for 0.001 µg/mL stimulant | -5.2 [-59.3 to 0.8] | -4.0 [-43.7 to 3.6] | 1.6 [-2.2 to 39.6]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported through the end of the study.
Description: Other [Not Including Serious] Adverse Events in the Untreated Control Arm were reported only in the 72 hours after any study-specific blood draws.
Groups:
- Placebo for Omalizumab/Milk OIT: Placebo for omalizumab: Placebo for omalizumab is injected subcutaneously every 2-4 weeks for 16 months at a volume designed to match that of the omalizumab treatment group (determined by the participant's IgE level and weight).
Arm/Group | Omalizumab/Milk OIT | Placebo for Omalizumab/Milk OIT | Untreated Control
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/29 | 1/20
Other Adverse Events (participants affected / at risk) | 26/28 | 28/29 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab/Milk OIT (N=28) | Placebo for Omalizumab/Milk OIT (N=29) | Untreated Control (N=20)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Omalizumab/Milk OIT (N=28) | Placebo for Omalizumab/Milk OIT (N=29) | Untreated Control (N=20)
Ear Pruritus (Ear and labyrinth disorders) | 1/27 (1) | 3/28 (102) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 3/27 (3) | 6/28 (11) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1/27 (1) | 2/28 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 12/27 (112) | 25/28 (531) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0/27 (0) | 2/28 (38) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3/27 (12) | 8/28 (21) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5/27 (10) | 3/28 (7) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2/27 (4) | 5/28 (75) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0/27 (0) | 2/28 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2/27 (12) | 6/28 (9) | 0 (0)
Oral Disorder (Gastrointestinal disorders) | 19/27 (373) | 27/28 (2441) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7/27 (21) | 11/28 (20) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 9 (11) | 0 (0)
Chest Discomfort (General disorders) | 3/27 (6) | 16/28 (225) | 0 (0)
Chest Pain (General disorders) | 2/27 (3) | 4/28 (7) | 0 (0)
Feeling Abnormal (General disorders) | 0/27 (0) | 2/28 (2) | 0 (0)
Sensation of foreign body (General disorders) | 0/27 (0) | 2/28 (2) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Ear Infection (Infections and infestations) | 3 (6) | 4 (5) | 0 (0)
Furuncle (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (6) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 9 (14) | 10 (13) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 7 (8) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 6 (8) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 5 (7) | 4 (6) | 0 (0)
Sinusitis (Infections and infestations) | 7 (11) | 5 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (17) | 12 (22) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (9) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0/27 (0) | 2/28 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0/27 (0) | 2/28 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (15) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/27 (11) | 14/28 (149) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/27 (0) | 2/28 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/27 (3) | 10/28 (43) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 11/27 (85) | 22/28 (202) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/27 (0) | 2/28 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6/27 (12) | 15/28 (102) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6/27 (15) | 22/28 (155) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2/27 (2) | 9/28 (12) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3/27 (5) | 12/28 (28) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10/27 (28) | 20/28 (264) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0/27 (0) | 5/28 (34) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 8/27 (47) | 23/28 (167) | 0 (0)
Flushing (Vascular disorders) | 4/27 (5) | 16/28 (92) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No